CLINICAL TRIAL: NCT06446791
Title: The Lateral Approach of the Webbed Neck: Mehri Turki Surgical Technique
Brief Title: Mehri Turki Surgical Technique of the Webbed Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Tahar Maamouri University Hospital (Other)
Responsible Party: Principal Investigator, Imen Turki Mehri, MD, Maxillofacial and aesthetic surgeon, Mohamed Tahar Maamouri University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Hospital MT Maamouri
Record Dates: First submitted 2024-05-24; First posted 2024-06-06 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Congenital Webbing of Neck
Keywords: Congenital abnormalities; Webbed neck; Surgical technique; Turner syndrome; Fetal cystic hygroma; Nuchal fold
MeSH Terms: conditions — Congenital Abnormalities; Turner Syndrome; Nuchal bleb, familial

STUDY DESIGN:
Intervention Model Description: Girls with congenital webbed neck deformity underwent the same surgical technique.
  Outcomes were analysed with long-term follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm interventionnal study (Other): A lateral approach surgical technique for the treatment of the webbed neck.
  Interventions: Procedure: Mehri Turki Surgical Technique of the Webbed Neck

INTERVENTIONS:
Procedure: Mehri Turki Surgical Technique of the Webbed Neck — The incision was made at the junction of the hairless skin and the hairy skin from the mastoid up to the acromion. A subcutaneous undermining allows direct visual control to excise the fibrotic band. Then the hairy skin with a triangular shape was excised. The closure of the defect was done after undermining an anterior cervical flap which was translated in a posterosuperior direction. Z plasty was performed in front of the acromion to prevent scar contracture. Surgical scars are concealed in the hairline which was well placed. The same procedure is done at the same surgical field on the other side to achieve perfect symmetry.
  Other Names: Mehri Turki Lateral approach Technique for the webbed beck

SUMMARY:
The webbed neck is one of the conspicuous deformities of Turner syndrome that presents a surgical challenge. Despite the availability of surgical techniques, surgical outcomes are not always acceptable and recurrence occurs. Mehri Turki performed a surgical technique based on a latéral cervical approach allowing direct visual control to manage the fibrotic band. It provides a high level of visual control so that vulnerable anatomic structures are easily protected.

DETAILED DESCRIPTION:
Five girls between 17 and 19 years old, with Turner syndrome, had a webbed neck (pterygium colli) with low and laterally displaced nuchal hairline. The surgical technique aims to correct neck contour and hairline placement while concealing cervical scars. Thus, Preoperative drawing delimitated the harmful triangular hairy skin next to the fibrous band extending from the mastoid to the acromion. Besides, the predefined design drawings provide the exact placement of the future hairline. Choosing a prone position for bilateral and symmetrical repair, the surgical technique was as follows:

The incision was made at the junction of the hairless skin and the hairy skin from the mastoid up to the lower end of the webbing skin, in front of the acromion and completed by Z plasty to avoid scar contracture. The subcutaneous skin was undermined in the anterolateral direction, exposing the fibrous fascial band which must be excised to prevent recurrence. the harmful skin having a triangular shape was excised considering the future hairline. Skin closure was done after the superior traction of the posterior cervical advancement.

ELIGIBILITY:
Inclusion Criteria:

* webbed neck with abnormal hairline

Exclusion Criteria:

* Surgical contraindication for any health concern
* Puberty age

Ages: 17 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01-27 (Actual); Primary Completion 2015-11-22 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Neck contour | Just at the postoperative outcome up to 24 months of follow-up
  Number of patient obtaining a normal neck contour without lateral fold
Posterior hairline placement | Just at the postoperative outcome up to 24 months of follow-up
  Number of patients with posterior hairline assent
Scars placement | Just at the postoperative outcome up to 24 months of follow-up
  Number of patients with a placement of scars at the level of the hairline

SECONDARY OUTCOMES:
Scars quality | from 8 months up to 24 months
  Scars evaluation according to Vancoover scare scale (VSS) for all patients The quality of post-operative scar was evaluated according to VSS as follows: combinations of 4 criteria (1) height (Normal/ 0; 0-2mm/ 1; 2-5mm/ 2 ; > 5mm / 3) and (2) pliability (Normal 0/ Supple 1/ Yielding 2/ Firm :3 Banding/4, Contracture/5); (3) Pigmentation (Normal : 0/ Hypopigmentation/ 1 Hyperpigmentation/ 2), and (4) Vascularity (Normal/0 Pink/ 1 Red/ 2 Purple/3).
  scars quality was judged as follows : Excellent result VSS <1 / Acceptable 1< VSS <5 ; Poor scar >5
Recurrece of the fold | 24 months
  Number of patients in whom the fold of the neck recurred

CONTACTS AND LOCATIONS:
Overall Officials: Imen Mehri Turki, Principal Investigator — University Hospital Mohamed Tahar Maamouri. Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mehri Turki I. Surgical correction of the webbed neck: an alternative lateral approach. GMS Interdiscip Plast Reconstr Surg DGPW. 2017 Mar 2;6:Doc04. doi: 10.3205/iprs000106. eCollection 2017. PMID 28275532
- [Result] Turki IM. Surgical techniques for the webbed neck: a narrative review with a comparative study and surgical decision-making algorithm for an optimal aesthetic result. Oral Maxillofac Surg. 2024 Jun;28(2):469-484. doi: 10.1007/s10006-023-01166-2. Epub 2023 Jun 20. PMID 37340235
- See also: Turki IM. Surgical techniques for the webbed neck: a narrative review with a comparative study and surgical decision-making algorithm for an optimal aesthetic result. Oral Maxillofac Surg. 2023 — https://link.springer.com/article/10.1007/s10006-023-01166-2
- See also: Mehri Turki I. Surgical correction of the webbed neck: an alternative lateral approach. GMS Interdiscip Plast Reconstr Surg DGPW. 2017 — https://www.egms.de/static/en/journals/iprs/2017-6/iprs000106.shtml